CLINICAL TRIAL: NCT01281397
Title: Bleeding Prediction in Patients Undergoing Cardiac Surgery Using Whole Blood Impedance Aggregometry and Rotational Thromboelastometry
Brief Title: Bleeding Prediction in Patients Following Cardiac Surgery Using Whole Blood Aggregometry and Thromboelastometry
Status: Terminated | Type: Observational
Why Stopped: After 148 patients enrolled, interim analysis revealed positive results in regard to primary hypothesis.
Sponsor: University of Zagreb (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other); Ministry of Science, Education and Sport, Republic of Croatia (Other Government)
Responsible Party: Principal Investigator, Petricevic Mate, Mate Petricevic M.D. , Ph.D., University of Zagreb
Other Study IDs: Project code: 198-1980976-097
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Heart Disease; Coronary Artery Disease; Aortic Valve Disease; Mitral Valve Disease
Keywords: cardiac surgery; aggregometry; thromboelastometry; platelet function; bleeding; antiplatelet therapy
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease; Aortic Valve Disease; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing elective cardiac surgery: Patients undergoing elective cardiac surgery will be enrolled in study. Data about antiplatelet therapy ingestion prior to surgery will be included.

SUMMARY:
Use of whole blood impedance aggregometry and rotational thromboelastometry can reveal useful data about platelet function and viscoelastic properties of blood clot in patients undergoing cardiac surgery.

The purpose of this study is to clarify whether it is possible to predict patients on excessive risk of perioperative bleeding using whole blood impedance aggregometry and rotational thromoelastometry.

Antiplatelet therapy is the cornerstone in treatment of patients with coronary artery disease. Another research goal is to determine the degree of response to antiplatelet therapy before and after surgery and to investigate whether patients by level of response to antiplatelet therapy before surgery have a higher risk of perioperative bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old
2. Elective cardiac surgery patients
3. Coronary artery disease
4. Aortic valve disease
5. Mitral valve disease
6. Ascendent aorta aneurysm
7. Combine coronary and valve disease
8. Cardiac surgery procedures using cardiopulmonary bypass

Exclusion Criteria:

1. Missing consent
2. Patients with emergent cardiac surgical procedures
3. Patients on antiplatelet therapy other than aspirin or clopidogrel
4. Patients with inaccurate antiplatelet therapy administration documentation
5. Missing data
6. Off-pump procedures
7. Patients younger than 18 years old
8. Patients with severe mental disorders
9. Intrinsic coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing elective cardiac surgery with cardiopulmonary bypass are enrolled in study.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Chest tube output in first 24 hours | 24 hours after surgical procedure

SECONDARY OUTCOMES:
Allogenic blood products transfusion | 7 days after surgery including the day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mate Petricevic, M.D., Principal Investigator — University hospital center Zagreb- Rebro; Bojan Biocina, M.D., Ph.D., Study Chair — University hospital center Zagreb - Rebro
Locations (1):
- University hospital center Zagreb- Rebro, Zagreb, Croatia, Croatia

REFERENCES:
- [Derived] Petricevic M, Biocina B, Milicic D, Svetina L, Boban M, Lekic A, Konosic S, Milosevic M, Gasparovic H. Activated coagulation time vs. intrinsically activated modified rotational thromboelastometry in assessment of hemostatic disturbances and blood loss after protamine administration in elective cardiac surgery: analysis from the clinical trial (NCT01281397). J Cardiothorac Surg. 2014 Sep 17;9:129. doi: 10.1186/1749-8090-9-129. PMID 25231271